CLINICAL TRIAL: NCT04398147
Title: A Randomized, Observer-Blind, Dose-escalation Phase I/II Clinical Trial of Ad5-nCoV Vaccine in Healthy Adults From 18 to <85 Years of Age in Canada
Brief Title: Phase I/II Clinical Trial of Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) in Canada
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Beijing Institute of Biotechnology (Other); Canadian Center for Vaccinology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ad5-nCoV-2020003
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: COVID-19; vaccine; Ad5; Safety; Immunogenicity; Dose-escalation; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Alzheimer Disease 5

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (28):
- phase ⅠLow single dose (18-<55) (Experimental): 12 subjects, Ad5-nCoV containing 5E10 vp, single dose, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- phase ⅠPlacebo low single dose (18-<55) (Placebo Comparator): 6 subjects, Placebo containing 0 vp, single dose, Intramuscular administration
  Interventions: Biological: Placebo
- phase ⅠLow 2 dose (18-<55) (Experimental): 12 subjects, Ad5-nCoV containing 5E10 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- phase ⅠPlacebo low 2 dose (18-<55) (Placebo Comparator): 6 subjects, Placebo containing 0 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Placebo
- phase ⅠLow single dose (65-<85) (Experimental): 12 subjects, Ad5-nCoV containing 5E10 vp, single dose, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- phase ⅠPlacebo low single dose (65-<85) (Placebo Comparator): 3 subjects, Placebo containing 0 vp, single dose, Intramuscular administration
  Interventions: Biological: Placebo
- phase ⅠLow 2 dose (65-<85) (Experimental): 12 subjects, Ad5-nCoV containing 5E10 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- phase ⅠPlacebo low 2 dose (65-<85) (Placebo Comparator): 3 subjects, Placebo containing 0 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Placebo
- phase ⅠMedium single dose (65-<85) (Experimental): 12 subjects, Ad5-nCoV containing 10E10 vp, single dose, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- phase ⅠPlacebo medium single dose (65-<85) (Placebo Comparator): 3 subjects, Placebo containing 0 vp, single dose, Intramuscular administration
  Interventions: Biological: Placebo
- phase ⅠMedium 2 dose (65-<85) (Experimental): 12 subjects, Ad5-nCoV containing 10E10 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- phase ⅠPlacebo medium 2 dose (65-<85) (Placebo Comparator): 3 subjects, Placebo containing 0 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Placebo
- Phase II Low single dose (18-<55) (Experimental): 50 subjects, Ad5-nCoV containing 5E10 vp, single dose, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- Phase II placebo low single dose (18-<55) (Placebo Comparator): 10 subjects，Placebo containing 0 vp, single dose, Intramuscular administration
  Interventions: Biological: Placebo
- Phase II Low 2 dose (18-<55) (Experimental): 50 subjects, Ad5-nCoV containing 5E10 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- Phase II placebo low 2 dose (18-<55) (Placebo Comparator): 10 subjects，Placebo containing 0 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Placebo
- Phase II Low single dose (55-<85) (Experimental): 50 subjects, Ad5-nCoV containing 5E10 vp, single dose, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- Phase II placebo low single dose (55-<85) (Placebo Comparator): 10 subjects，Placebo containing 0 vp, single dose, Intramuscular administration
  Interventions: Biological: Placebo
- Phase II Low 2 dose (55-<85) (Experimental): 50 subjects, Ad5-nCoV containing 5E10 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- Phase II placebo low 2 dose (55-<85) (Placebo Comparator): 10 subjects，Placebo containing 0 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Placebo
- Phase II medium single dose (55-<85) (Experimental): 50 subjects, Ad5-nCoV containing 10E10 vp, single dose, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- Phase II placebo medium single dose (55-<85) (Placebo Comparator): 10 subjects，Placebo containing 0 vp, single dose, Intramuscular administration
  Interventions: Biological: Placebo
- Phase II medium 2 dose (55-<85) (Experimental): 50 subjects，Ad5-nCoV containing 10E10 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- Phase II placebo medium 2 dose (55-<85) (Placebo Comparator): 10 subjects，Placebo containing 0 vp, 2 dose 56 days apart, Intramuscular administration
  Interventions: Biological: Placebo
- Phase II Low 1 or 2 dose (18-<55) (Experimental): 100 subjects，Ad5-nCoV containing 5E10 vp, 1or2 dose, Intramuscular administration ，according to the Previous trial results
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- Phase II placebo 1 or 2 dose (18-<55) (Placebo Comparator): 20 subjects，placebo containing 0 vp, 1or2 dose, Intramuscular administration
  Interventions: Biological: Placebo
- Phase II Low or medium dosage 1 or 2 dose (55-<85) (Experimental): 100 subjects，Ad5-nCoV containing 5E10 vp or 10E10vp, 1or2 dose, Intramuscular administration，according to the Previous trial results
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- Phase II placebo Low or medium,1 or 2 dose (55-<85) (Placebo Comparator): 20 subjects，placebo containing 0 vp, 1or2 dose, Intramuscular administration
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) — Intramuscular administration
  Arms: Phase II Low 1 or 2 dose (18-<55); Phase II Low 2 dose (18-<55); Phase II Low 2 dose (55-<85); Phase II Low or medium dosage 1 or 2 dose (55-<85); Phase II Low single dose (18-<55); Phase II Low single dose (55-<85); Phase II medium 2 dose (55-<85); Phase II medium single dose (55-<85); phase ⅠLow 2 dose (18-<55); phase ⅠLow 2 dose (65-<85); phase ⅠLow single dose (18-<55); phase ⅠLow single dose (65-<85); phase ⅠMedium 2 dose (65-<85); phase ⅠMedium single dose (65-<85)
Biological: Placebo — Intramuscular administration
  Arms: Phase II placebo 1 or 2 dose (18-<55); Phase II placebo Low or medium,1 or 2 dose (55-<85); Phase II placebo low 2 dose (18-<55); Phase II placebo low 2 dose (55-<85); Phase II placebo low single dose (18-<55); Phase II placebo low single dose (55-<85); Phase II placebo medium 2 dose (55-<85); Phase II placebo medium single dose (55-<85); phase ⅠPlacebo low 2 dose (18-<55); phase ⅠPlacebo low 2 dose (65-<85); phase ⅠPlacebo low single dose (18-<55); phase ⅠPlacebo low single dose (65-<85); phase ⅠPlacebo medium 2 dose (65-<85); phase ⅠPlacebo medium single dose (65-<85)

SUMMARY:
This study is a phase I /II adaptive clinical trial to evaluate the safety, tolerability and the Immunogenicity of Ad5-nCoV in healthy adults from 18 to <55 and 65 to <85 years of age，with the randomized, observer-blind, dose-escalation design

DETAILED DESCRIPTION:
A total of 96 healthy adult volunteers will be vaccinated in phase I stepwised according to the dose-escalation design from the younger adults(18 to <55) to the older adults(65 to <85). There are 2 dosage level used in this phase: 5E10vp and 10E10vp, and 2 dose schedules: single dose and 2 dose. According to the pre-defined adaptive design standards, the trial will moved from Phase I to Phase II. In the phase II portion, A total of 600 healthy adult volunteers will be vaccinated according to the dose-escalation design from the younger adults(18 to <55) to the older adults(55 to <85). There are 2 dosage levels and schedules used in this phase，and will determine a final dose and schedule by the end. Some cohorts in the phase II trial will be included in the subsequent phase III trial.

ELIGIBILITY:
Inclusion criteria for the phase I portion of the study:

* Healthy adults from 18 to <55 and 65-<85 years of age at the time of enrollment;
* Able to provide consent to participate in and having signed an Informed Consent Form (ICF);
* Able and willing to complete all the scheduled study procedures during the whole study follow-up period (about 6-8 months, depending on group);
* Negative result of HIV, hepatitis B and C screening;
* Oral temperature < 38.0℃;
* Negative IgG and IgM antibodies against COVID-19;
* Negative result of real-time quantitative PCR screening of nasopharyngeal swabs/sputum for SARS-CoV-2;
* A body mass index (BMI) between 18-35;
* Hematological examination is within normal range, or no greater than a grade 1 abnormality and no clinical significance as assessed by the study investigator (including white blood cell count, lymphocyte count, neutrophil count, eosinophil count, platelet, hemoglobin, alanine aminotransferase ALT, aspartate aminotransferase AST, total bilirubin, blood glucose and creatinine);
* Transient mild laboratory abnormalities may be rescreened once and the participant will be deemed eligible if the laboratory repeat test is normal as per local laboratory normal values and investigator assessment.
* Good general health status, as determined by history and physical examination no greater than 14 days prior to administration of the test article.
* If female of child-bearing potential and heterosexually active, has practiced adequate contraception for 30 days prior to injection, has a negative pregnancy test on the day of injection, and has agreed to continue adequate contraception until 180 days after injection. (Please refer to the glossary for the definition of child-bearing potential and adequate contraception).

Inclusion criteria for the phase II portion of the study will be detailed in an amended synopsis/study protocol.

Exclusion criteria for the phase I portion of the study:

* Personal history of seizure disorder, encephalopathy or psychosis;
* Allergic history to any vaccine, or allergic to any ingredient of the Ad5-nCoV;
* Woman is pregnant or lactating, positive urine pregnancy test or plan to become pregnant during the next 6 months;
* Any acute febrile disease (oral temperature ≥38.0℃ or active infectious disease on the day of vaccination;
* Medical history of SARS (SARS-CoV-1);
* Serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension not controlled with medication;
* Serious chronic disease such as asthma, diabetes and thyroid disease, etc.;
* Congenital or acquired angioedema;
* Immunodeficiency, asplenia or functional asplenia;
* Platelet disorder or other bleeding disorder that may cause intramuscular injection contraindication;
* Immunosuppressive medication, anti-allergic, cytotoxic therapy, inhaled corticosteroids (excluding corticosteroid spray for allergic rhinitis, surface corticosteroid therapy for acute non-complicated dermatitis) in the last 6 months;
* Prior administration of blood products in last 4 months;
* Other vaccination(s) or investigational drugs within 1 month before study onset, or planned use during the study period;
* Prior administration of live attenuated vaccine within 1 month before study onset;
* Prior administration of subunit or inactivated vaccine within 14 days before study onset;
* Current anti-tuberculosis therapy;
* Any condition that in the opinion of the investigators may interfere with the participants' compliance or evaluation of study objectives or informed consent (i.e. medical, psychological, social or other conditions, etc.) Exclusion criteria for the phase II portion of the study will be detailed in an amended synopsis/study protocol.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 696 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of the Solicited AE in all groups | 0-6 days after each vaccination
  The occurrence of Solicited AE in all groups within 0-6 days after each vaccination;
Incidence of Unsolicited AE in all groups | 0-28 days after each vaccination
  The occurrence of Unsolicited AE in all groups within 0-28 days after each vaccination.
Incidence of Serious adverse events (SAE) in all groups | 6 months after the final vaccination
  The occurrence of Serious adverse events (SAE) in all groups within 6 months after the final vaccination.

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of the IgG antibody against SARS-CoV-2 (ELISA method); | Day 0, Day 14, Day 28, Day 84 and Day 168 after vaccination in the one dose group and Day 0, 14, 28, 56, 70, 84, and 224 in the two dose group
  Geometric mean titer (GMT) of the IgG antibody against SARS-CoV-2 measured on Day 0, Day 14, Day 28, Day 84 and Day 168 after vaccination in the one dose group and Day 0, 14, 28, 56, 70, 84, and 224 in the two dose group (ELISA method);
Seroconversion rate of the IgG antibody against SARS-CoV-2(ELISA method ) | Day 14, Day 28, Day 84 and Day 168 after vaccination in the one dose group and Day 14, 28, 56, 70, 84, and 224 in the two dose group
  Seroconversion rate (%of subjects with 4-fold or greater increase in antibody level) of the IgG antibody against SARS-CoV-2 measured on Day 14, Day 28, Day 84 and Day 168 after vaccination in the one dose group and Day 14, 28, 56, 70, 84, and 224 in the two dose group (ELISA method );
Geometric Mean Increase Ratio (GMI) of the specific antibody against SARS-CoV-2(ELISA method); | Day 14, Day 28, Day 84 and Day 168 after vaccination in the one dose group and Day 14, 28, 56, 70, 84, and 224 in the two dose group
  Geometric Mean Increase Ratio (GMI) of the specific antibody against SARS-CoV-2 measured on Day 14, Day 28, Day 84 and Day 168 after vaccination in the one dose group and Day 14, 28, 56, 70, 84, and 224 in the two dose group (ELISA method);
Geometric mean titer (GMT) of the neutralizing antibody against SARS-CoV-2(Pseudo-viral neutralization assay) | Day 0, Day 14, Day 28 and Day 168 after vaccination in the one dose group and Day 0, 14, 28, 56, 70, 84, and 224 in the two dose group
  Geometric mean titer (GMT) of the neutralizing antibody against SARS-CoV-2 measured on Day 0, Day 14, Day 28 and Day 168 after vaccination in the one dose group and Day 0, 14, 28, 56, 70, 84, and 224 in the two dose group (Pseudo-viral neutralization assay)
Seroconversion rate of the neutralizing antibody against SARS-CoV-2(Pseudo-viral neutralization assay) | Day 14, Day 28 and Day 168 after vaccination in the one dose group and Day 14, 28, 56, 70, 84, and 224 in the two dose group
  Seroconversion rate of the neutralizing antibody against SARS-CoV-2 measured on Day 14, Day 28 and Day 168 after vaccination in the one dose group and Day 14, 28, 56, 70, 84, and 224 in the two dose group(Pseudo-viral neutralization assay);
Geometric mean increase ratio (GMI) of neutralizing antibody against SARS-CoV-2 (Pseudo-viral neutralization assay) | Day 14, Day 28 and Day 168 after vaccination in the one dose group and Day 14, 28, 56, 70, 84, and 224 in the two dose group
  Geometric mean increase ratio (GMI) of neutralizing antibody against SARS-CoV-2 measured on Day 14, Day 28 and Day 168 after vaccination in the one dose group and Day 14, 28, 56, 70, 84, and 224 in the two dose group (Pseudo-viral neutralization assay)
Geometric Mean Titer (GMT) of the neutralizing antibody against adenovirus type 5 vector | Day 0, Day 14, Day 28, Day 84 and Day 168 after vaccination in the one dose group and Day 0, 14, 28, 56, 70, 84, and 224 in the two dose group
  Geometric Mean Titer (GMT) of the neutralizing antibody against adenovirus type 5 vector measured on Day 0, Day 14, Day 28, Day 84 and Day 168 after vaccination in the one dose group and Day 0, 14, 28, 56, 70, 84, and 224 in the two dose group;
Geometric mean increase ratio (GMI) of the neutralizing antibody against adenovirus type 5 vector | Day 14, Day 28, Day 84 and Day 168 after vaccination in the one dose group and Day 14, 28, 56, 70, 84, and 224 in the two dose group
  Geometric mean increase ratio (GMI) of the neutralizing antibody against adenovirus type 5 vector measured on Day 14, Day 28, Day 84 and Day 168 after vaccination in the one dose group and Day 14, 28, 56, 70, 84, and 224 in the two dose group
cellular immune response by ELISpot | on Day 0, Day 14, Day 28 and Day 168 in the one dose group and Day 0, 14, 28, 56, 70, 84, and 224 in the two dose group
  The positive rate of IFN-γ stimulated by S protein overlapping peptide library detected by ELISpot
cellular immune response by ICS | Day 0, Day 14, Day 28 and Day 168 in the one dose group and Day 0, 14, 28, 56, 70, 84, and 224 in the two dose group
  The positive rate of IFN-γ, TNF-α, and IL-2 expressed by CD4+ and CD8+ T lymphocytes stimulated by S protein overlapping peptide library detected by Intracellular Cytokine Staining (ICS);

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Halperin, MD, Principal Investigator — Canadian Center for Vaccinology; Joanne M Langley, MD, Principal Investigator — Canadian Center for Vaccinology
Locations (1):
- Canadian Center for Vaccinology, Halifax, Canada

IPD SHARING:
Plan to Share IPD: No